CLINICAL TRIAL: NCT04808505
Title: An Open-label Study to Evaluate the Safety, Efficacy, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Cipaglucosidase Alfa/Miglustat in Both ERT-experienced and ERT-naïve Pediatric Subjects With Infantile-onset Pompe Disease Aged 0 to < 18 Years
Brief Title: A Study to Evaluate the Safety, Efficacy, PK, PD and Immunogenicity of Cipaglucosidase Alfa/Miglustat in IOPD Subjects Aged 0 to <18
Acronym: ROSSELLA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATB200-08
Expanded Access: NCT04327973 (Available)
Record Dates: First submitted 2021-03-10; First posted 2021-03-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Glycogen Storage Disease Type II Infantile Onset
MeSH Terms: interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Cipaglucosidase Alfa/Miglustat in ERT-experienced pediatric IOPD subjects (Experimental): Pediatric IOPD subjects 6 months to <18 years experiencing clinical decline
  Interventions: Biological: Cipaglucosidase alfa; Drug: Miglustat
- Cohort 2: Cipaglucosidase Alfa/Miglustat in ERT-naïve pediatric IOPD subjects (Experimental): Pediatric IOPD subjects <6 months
  Interventions: Biological: Cipaglucosidase alfa; Drug: Miglustat

INTERVENTIONS:
Biological: Cipaglucosidase alfa — Sterile lyophilized powder intravenous (IV) infusion
  Other Names: ATB200
Drug: Miglustat — 65 mg oral capsules
  Other Names: AT2221

SUMMARY:
This is a Phase 3, open-label, multicenter study to evaluate the safety, efficacy, PK, PD, and immunogenicity of cipaglucosidase alfa/miglustat treatment in ERT-experienced and ERT-naïve pediatric subjects with IOPD.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

1. Male or female subjects who are aged 6 months to < 18 years on Day 1
2. Subject must have documentation of IOPD genotype
3. Subject must have had hypertrophic cardiomyopathy at the time of diagnosis
4. Subject must have received ERT for at least 6 months immediately before enrollment. For subjects whose ERT dosage has been modified, the subject must have been on the modified dosage and regimen for at least 3 months before enrollment
5. Subjects aged ≥ 12 to < 18 years must perform one valid 6-minute walk test (6MWT) (≥ 75 meters) at screening; Subjects aged ≥ 5 to < 12 years must perform one valid 6MWT (≥ 40 meters) at screening; Subjects aged 18 months to < 5 years must be ambulatory and assessed to be likely to be able to perform 6MWT (≥ 40 meters) when they turn 5 years old
6. Subjects must have experienced a clinical decline on their current rhGAA dose and frequency

Cohort 2:

1. Male or female subjects who are aged 0 to <6 months at Day 1
2. Subject must have documentation of IOPD genotype
3. Subject must have had hypertrophic cardiomyopathy at the time of diagnosis
4. Subject is ERT-naïve

Long-term Extension (Cohort 1 or Cohort 2):

1. Subject must have, in the opinion of the investigator, benefited from therapy with cipaglucosidase alfa/miglustat during the 104-week primary treatment period with no significant safety concerns.

Exclusion Criteria:

Cohort 1 and Cohort 2, unless specified

1. Subject requires invasive ventilation (eg, tracheostomy)
2. Subject is CRIM negative and has not received prophylactic immunomodulation (Cohort 1); Subject is CRIM negative and will not be receiving prophylactic immunomodulation (Cohort 2)
3. Subject has a history of life-threatening IARs/hypersensitivity (eg, anaphylaxis and severe cutaneous reactions) to ERT (eg, alglucosidase alfa, cipaglucosidase alfa, miglustat) or other iminosugars, or to any of the excipients, where rechallenge was unsuccessful
4. Subject has prior history of illness or condition known to affect motor function
5. Female subject is pregnant (or intends to get pregnant) or breastfeeding at screening (Cohort 1)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with infusion-associated reactions (IARs) | 104 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - University of Florida Clinical Research Center, Gainesville, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Duke University Early Phase Research Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Clinical and Translational Sciences Institute, Salt Lake City, Utah
- Germany (4):
  - Universitätsklinikum Gießen und Marburg GmbH, Zentrum fur Kinderheilkunde und Jugendmedizin Abteilung fur Kinderneurologic, Sozialpadiatric und Epileptologie, Giessen
  - Universitätsklinikum Heidelberg - Pädiatrisches Klinisch-Pharmakologisches Studienzentrum (paedKliPS), Heidelberg
  - SphinCS GmbH, Höchheim
  - Universitätsklinikum Münster Klinik für Kinder- und Jugendmedizin Albert-Schweitzer-Campus 1, Münster
- AOU Federico II, Naples, Italy
- Erasmus MC, Sophia Kinderziekenhuis, Rotterdam, Netherlands
- National Taiwan University Hospital, Taipei, Taiwan
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No